CLINICAL TRIAL: NCT05875467
Title: Evaluation of Prototype Game for Simulation for Environmental Exposure Education
Brief Title: Evaluation of Prototype for Simulation for Environmental Exposure Education (SE3)
Acronym: SE3
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: dfusion Inc (Industry)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R43ES024563; 1R43ES034563-01 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Effect of Game in Increasing Environmental Health Literacy
Keywords: environmental health; game; air quality; STEM; health literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm, Intervention with SE3 Game (Experimental): This is a single arm study. This arm will receive the intervention. This intervention is a prototype of online game, about 50 minutes in duration. The online game provides gameplay that allows the user, with a gameplay narrative, to identify and remove sources of environmental hazards in the home environment. Participants play the prototype game for about 50 minutes at which time the intervention is complete.
  Interventions: Other: SE3 Game

INTERVENTIONS:
Other: SE3 Game — A prototype online game designed to increase environmental health literacy

SUMMARY:
The goal of this clinical trial is to test a prototype of a new educational game about environmental health literacy with middle school age youth. The main questions it aims to answer are:

* Does playing the game increase knowledge about environmental health?
* Does playing the game improve environmental health literacy?
* Does playing the game increase interest and confidence in science?

Participants will be asked to:

* Take a survey at the beginning of the study
* Play the game for a minimum of 50 minutes
* Take a survey at the end of the study

DETAILED DESCRIPTION:
The proposed project will establish the technical merit and feasibility of producing and using a serious game to improve environmental health literacy among young people. A small evaluation is being conducted to assess the impact of the prototype game on environmental health knowledge, literacy, ability to understand mitigation, and impact on science interest and confidence.

Participants will be middle school youth, typically ages 11-15, who are currently enrolled in middle school. Participants are being recruited by the projects education advisor (CA) and youth community board members (MI).

Investigators will conduct an evaluation with 45 middle school age participants from communities disproportionately impacted by environmental risk. The goal is to test the usability and playability of the prototype and assess the games impact on outcomes. The participant will complete a short online pre-test assessment (environmental health knowledge), participate in either a 50 play session or a week long play period logging a minimum of 50 minutes. At the end of the play period the participant will complete a short post-test with similar questions to the pre-test plus additional questions about their usage, satisfaction with, and enjoyment of the game. During independent game use, the app will collect metrics on usage, player performance, and conditional knowledge including the ability to apply concepts in context. Participants will each receive a $100 gift card.

ELIGIBILITY:
Inclusion Criteria:

* In middle school.
* Ability to use a mobile tablet.
* Have access to wifi in location of intervention implementation.
* Reside in the geographic areas of implementation: California, Michigan, Florida

Exclusion Criteria:

* Age not within middle school range.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Kuhn, MA, Principal Investigator — dfusion Inc
Locations (2):
- United States (2):
  - Monroe Middle School, San Jose, California
  - Virtual Study, Scotts Valley, California

IPD SHARING:
Plan to Share IPD: No
The research is being conducted under a Small Business Innovation Grant (SBIR) in support of product development and is considered proprietary to the business.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place during an approximately one-month period. Participants were recruited in one middle-school classroom (two classes) in San Jose, CA. Additional participants for across the country were recruited through referrals from teachers and other education advisors.
Pre-assignment Details: This was a single arm study so participants were not assigned to a group. No recruited participants were excluded prior to participation.
Period: Overall Study
Arm/Group | Single Arm, Intervention With SE3 Game
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm, Intervention With SE3 Game
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 13.6 [11 to 15]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 23
  Gender: Female | 26
  Gender: Non binary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 2
  White | 17
  More than one race | 16
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Environmental Health Indoor Air Pollution Knowledge Score
Description: Based on a scale created for this study the Environmental Health Indoor Air Pollution Knowledge Score is comprised of a series of questions about indoor environmental pollution. The scores from the question are summed to create a total score. The scale ranges from 0 to 17 with a higher score indicating greater knowledge.
Time Frame: Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm, Intervention With SE3 Game
Number analyzed (Participants) | 50
score on a scale | 1.38 (4.67)
Statistical Analysis 1: Comparison: Single Arm, Intervention With SE3 Game; Test type: Superiority; p = .042, t-test, 2 sided

2. Secondary Outcome: Change in Environmental Health Mitigation Knowledge Score
Description: Based on a scale created for this study the Environmental Mitigation Knowledge Score is comprised of a series of questions about what can mitigate indoor air pollution. The scores from the questions are summed to create a total score. The score range is 0 to 14 with higher scores indicating greater knowledge.
Time Frame: Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm, Intervention With SE3 Game
Number analyzed (Participants) | 50
score on a scale | 4.85 (1.75)
Statistical Analysis 1: Comparison: Single Arm, Intervention With SE3 Game; Test type: Superiority; p = .928, t-test, 2 sided

3. Secondary Outcome: Change in Environmental Health Interest Score
Description: Based on a scale created for this study the Environmental Health Interest Score is comprised of a series of questions to assess interest. The scores from the question are summed to create a total score. The score range is 4 to 24 with higher scores indicating greater environmental health literacy.
Time Frame: Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm, Intervention With SE3 Game
Number analyzed (Participants) | 50
score on a scale | .932 (2.59)
Statistical Analysis 1: Comparison: Single Arm, Intervention With SE3 Game; Test type: Superiority; p = .022, t-test, 2 sided

4. Secondary Outcome: Change in Science Interest and Confidence Score
Description: Based on a scale created for the Science Interest and Confidence Score is comprised of a series of questions about interest in science and perceived skill in science. The scores from the question are summed to create a total score. The score range is 1 to 5, with higher scores indicating more science interest and confidence.
Time Frame: Day 1 to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm, Intervention With SE3 Game
Number analyzed (Participants) | 50
score on a scale | 1.64 (3.57)
Statistical Analysis 1: Comparison: Single Arm, Intervention With SE3 Game; Test type: Superiority; p = .004, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From initial recruitment to post test was a 30 day period. Data were collected during this period.
Arm/Group | Single Arm, Intervention With SE3 Game
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT05875467/Prot_SAP_000.pdf